CLINICAL TRIAL: NCT06595108
Title: Atezolizumab and Bevacizumab With Stereotactic Body Radiotherapy for Advanced Hepatocellular Carcinoma
Acronym: A-BEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hwa Kyung Byun, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-2024-0026
Record Dates: First submitted 2024-07-29; First posted 2024-09-19 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Advanced Hepatocellular Carcinoma; Chemotherapy; Stereotactic Body Radiotherapy
Keywords: atezolizumab-bevacizumab; SBRT
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Patients with advanced hepatocellular carcinoma who are indicated for the first-line atezolizumab-bevacizumab combination chemotherapy should begin stereotactic body radiotherapy to one or more but not more than five sites for primary cancer and/or metastatic lesions.
Masking Description: Patients with advanced hepatocellular carcinoma who are indicated for the first-line atezolizumab-bevacizumab combination chemotherapy should begin stereotactic body radiotherapy to one or more but not more than five sites for primary cancer and/or metastatic lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced hepatocellular carcinoma (Experimental): Patients indicated for the first-line atezolizumab-bevacizumab combination therapy are the primary subjects, and those voluntarily agree to the clinical trial after explanation of the study, are enrolled in the study.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Patients with advanced hepatocellular carcinoma who are indicated for the first-line atezolizumab-bevacizumab combination therapy are the primary subjects, and they should begin stereotactic radiotherapy to one or more but not more than five sites for primary cancer and/or metastatic lesions within two month before and after the start date of atezolizumab-bevacizumab combination therapy.

SUMMARY:
To determine the efficacy and safety of atezolizumab-bevacizumab combination therapy plus stereotactic body radiotherapy(SBRT) in patients with advanced hepatocellular carcinoma, Subjects will start SBRT for one or more primary cancers and/or metastatic lesions and no more than 5 sites within two month before and after the start date of atezolizumab-bevacizumab combination therapy.

In this study, it is expected to improve the treatment response rate of atezolizumab-bevacizumab therapy, which is currently first-line chemotherapy but has a low treatment response rate.

DETAILED DESCRIPTION:
The subjects with advanced hepatocellular carcinoma who are indicated for the first-line atezolizumab-bevacizumab combination therapy are the primary subjects, and if they voluntarily agree to the clinical trial after explanation of the clinical trial, they are included in the clinical trial. Subjects should begin SBRT(stereotactic body radiotherapy) to one or more but not more than five sites for primary cancer and/or metastatic lesions within two month before and after the start date of atezolizumab-bevacizumab combination therapy.

The followings are evaluation items for each visit.

Visit 1 (-6~0 weeks) ± 7days *Screening

* Informed consent form
* Inclusion Criteria/ Exclusion Criteria
* Medical history and physical examination
* Staging via CT, MRI, PET-CT, etc. (PET-CT examination is not compulsory)
* CBC, SMA, PT/aPTT, Tumor markers, Biomarkers
* Stool microbiota NGS
* QoL Questionnaire(EORTC-QLQ-C30 V3)

Visit 2 (0~7 weeks) ± 7 days *During SBRT

* Confirmation of adverse events
* QoL Questionnaire(EORTC-QLQ-C30 V3)

Visit 3 (1~8 weeks) *1 week after SBRT

* Confirmation of adverse events
* CBC, SMA, PT/aPTT, Tumor markers, Biomarkers
* QoL Questionnaire(EORTC-QLQ-C30 V3)

Visit 4 (6~9 weeks) ± 7 days *After 2 cycles of chemotherapy

* Confirmation of adverse events
* CBC, SMA, PT/aPTT, Tumor markers, Biomarkers
* Stool microbiota NGS
* QoL Questionnaire(EORTC-QLQ-C30 V3)

Visit: 5~12 (3~36 months) ± 2 weeks *Follow-up

* Confirmation of adverse events
* Evaluation of effectiveness* (Imaging tests, Tumor markers, CBC, SMA, PT/aPTT are performed according to the need)
* QoL Questionnaire(EORTC-QLQ-C30 V3)

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 to 80 years old
2. Liver function Child-Pugh class A
3. ECOG 0-1
4. Patient clinically or pathologically diagnosed with hepatocellular carcinoma
5. Advanced hepatocellular carcinoma that is inoperable
6. Satisfies the dose limits for normal organs and lesions of an appropriate size to be included in the scope of radiotherapy.

Exclusion Criteria:

1. Brain metastases
2. Have a history of malignancy other than hepatocellular carcinoma within the last 5 years (except for malignancies with little risk of metastasis or death, e.g., adequately treated cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, tubular carcinoma in situ, or stage 1 uterine cancer.)
3. Subjects with a high probability of untreated gastric or esophageal varices or bleeding
4. Serious uncontrolled medical comorbidities
5. History of liver transplant surgery
6. Autoimmune liver disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 6 month | 6 months after registration
  The primary endpoint is to improve 6-month progression-free survival rate in the treatment group compared to those existing literature. Progression-free survival and overall survival are evaluated using the Kaplan-Meier curve. Verified through one sample proportion test.

SECONDARY OUTCOMES:
Overall survival | 36 months after registration
  Progression-free survival and overall survival are evaluated using the Kaplan-Meier curve. Verified through one sample proportion test.
Objective response rate | 36 months after registration
  Objective response rate will be ratepresented as a proportion of the total.
Adverse event (Toxicity) | 36 months after registration
  Toxicity will be evaluated using CTCAE version 5.0 and presented as a proportion of the total.
Tumor marker response: AFP, PIVKA-II | 36 months after registration
  Tumor markers and biological markers are descriptive as statistics such as mean, standard deviation, and median for continuous data will be presented, and changes in values before and after treatment will be compared and evaluated using paired t-test or Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Hwakyung BYUN, Phd, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng L, Xu J, Ye Y, Wang Y, Luo S, Gong X. The Combination of Radiotherapy With Immunotherapy and Potential Predictive Biomarkers for Treatment of Non-Small Cell Lung Cancer Patients. Front Immunol. 2021 Sep 21;12:723609. doi: 10.3389/fimmu.2021.723609. eCollection 2021. PMID 34621270
- [Background] Demaria S, Golden EB, Formenti SC. Role of Local Radiation Therapy in Cancer Immunotherapy. JAMA Oncol. 2015 Dec;1(9):1325-32. doi: 10.1001/jamaoncol.2015.2756. PMID 26270858
- [Background] Demaria S, Guha C, Schoenfeld J, Morris Z, Monjazeb A, Sikora A, Crittenden M, Shiao S, Khleif S, Gupta S, Formenti SC, Vikram B, Coleman CN, Ahmed MM. Radiation dose and fraction in immunotherapy: one-size regimen does not fit all settings, so how does one choose? J Immunother Cancer. 2021 Apr;9(4):e002038. doi: 10.1136/jitc-2020-002038. PMID 33827904
- [Background] Byun HK, Kim N, Park S, Seong J. Acute severe lymphopenia by radiotherapy is associated with reduced overall survival in hepatocellular carcinoma. Strahlenther Onkol. 2019 Nov;195(11):1007-1017. doi: 10.1007/s00066-019-01462-5. Epub 2019 Apr 15. PMID 30989242
- [Background] Theelen WSME, Peulen HMU, Lalezari F, van der Noort V, de Vries JF, Aerts JGJV, Dumoulin DW, Bahce I, Niemeijer AN, de Langen AJ, Monkhorst K, Baas P. Effect of Pembrolizumab After Stereotactic Body Radiotherapy vs Pembrolizumab Alone on Tumor Response in Patients With Advanced Non-Small Cell Lung Cancer: Results of the PEMBRO-RT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Sep 1;5(9):1276-1282. doi: 10.1001/jamaoncol.2019.1478. PMID 31294749
- [Background] Luke JJ, Lemons JM, Karrison TG, Pitroda SP, Melotek JM, Zha Y, Al-Hallaq HA, Arina A, Khodarev NN, Janisch L, Chang P, Patel JD, Fleming GF, Moroney J, Sharma MR, White JR, Ratain MJ, Gajewski TF, Weichselbaum RR, Chmura SJ. Safety and Clinical Activity of Pembrolizumab and Multisite Stereotactic Body Radiotherapy in Patients With Advanced Solid Tumors. J Clin Oncol. 2018 Jun 1;36(16):1611-1618. doi: 10.1200/JCO.2017.76.2229. Epub 2018 Feb 13. PMID 29437535
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Timmerman R. A Story of Hypofractionation and the Table on the Wall. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):4-21. doi: 10.1016/j.ijrobp.2021.09.027. No abstract available. PMID 34919882